CLINICAL TRIAL: NCT07160114
Title: Task-oriented Training With Electrical Stimulation Glove on Hand Function and Dexterity in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha waris, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0031
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Chronic Stroke Patient
Keywords: Stroke rehabilitation; Electrical stimulation glove; Task-oriented training; Upper extremity function; Hand dexterity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-Oriented Training with Electrical Stimulation Glove (Experimental): Participants receive task-oriented training combined with an electrical stimulation glove. Sessions include warm-up exercises, functional activities (such as pegboard tasks, grasp-and-release of objects, writing, and simulated daily activities), and cool-down stretches. The glove delivers low-intensity electrical impulses to the wrist and finger muscles during training to facilitate neuromuscular activation and enhance motor recovery. Sessions last approximately 60 minutes, three times per week for 8 weeks.
  Interventions: Device: Electrical Stimulation Glove with Task-Oriented Training
- Task-Oriented Training Only (Active Comparator): Participants receive task-oriented training without the electrical stimulation glove. Sessions include warm-up exercises, functional activities (such as pegboard placement, grasp-and-release of objects, writing or drawing, and simulated daily activities), and cool-down stretches. This protocol provides standard rehabilitation focusing on functional use of the affected hand. Sessions last approximately 60 minutes, three times per week for 8 weeks.
  Interventions: Behavioral: Task-Oriented Training Only

INTERVENTIONS:
Device: Electrical Stimulation Glove with Task-Oriented Training — Participants perform structured task-oriented training while wearing an electrical stimulation glove. The glove is embedded with electrodes that deliver low-intensity electrical impulses to the wrist and finger muscles during functional tasks. Training includes warm-up range of motion and stretching, 40 minutes of functional activities such as pegboard tasks, object manipulation, writing, and daily living tasks, followed by cool-down exercises. The intervention is delivered in 60-minute sessions, three times per week, for 8 weeks.
  Arms: Task-Oriented Training with Electrical Stimulation Glove
Behavioral: Task-Oriented Training Only — Participants receive task-oriented training without the electrical stimulation glove. Training includes warm-up range of motion and stretching, 40 minutes of functional activities such as pegboard placement, grasp-and-release, writing or drawing, and simulated daily living tasks, followed by cool-down exercises. The intervention is delivered in 60-minute sessions, three times per week, for 8 weeks.
  Arms: Task-Oriented Training Only

SUMMARY:
Stroke often causes long-lasting weakness and difficulty using the hands, which limits independence in daily life. Many patients find it hard to perform everyday tasks such as dressing, eating, or writing. Rehabilitation usually includes task-oriented training (TOT), which means practicing meaningful activities that mimic real-life situations.

This study is testing whether adding a new device called an electrical stimulation glove (ESG) can make hand training more effective for people living with chronic stroke. The glove delivers gentle electrical impulses to the muscles in the hand while patients practice functional tasks. This stimulation may help activate weak muscles and improve coordination during rehabilitation.

Participants in this study are divided into two groups:

One group receives task-oriented training with the electrical stimulation glove,

The other group receives task-oriented training only.

Therapy includes warm-up exercises, task practice such as pegboard activities, grasping and releasing objects, and everyday skills, followed by cool-down exercises.

The study is being carried out at CMH Multan, Pakistan, and involves adult men and women between 40 and 60 years of age who have experienced a stroke more than six months earlier. Outcomes are measured with standard rehabilitation tools that assess hand function, motor recovery, and dexterity.

This research may help determine whether the electrical stimulation glove can be used alongside routine rehabilitation programs to support better recovery of hand function in people with stroke.

DETAILED DESCRIPTION:
Background and Rationale Stroke is a major cause of long-term disability worldwide. Many stroke survivors experience chronic upper limb impairment, including weakness, stiffness, and reduced dexterity, which limits their ability to perform daily activities. Task-oriented training is a widely used rehabilitation approach that focuses on practicing functional, goal-directed movements to restore independence. Electrical stimulation has also been shown to support neuromuscular activation and promote neuroplasticity. Integrating these two strategies into a single wearable device - an electrical stimulation glove (ESG) - may offer a novel and affordable rehabilitation option.

Study Objectives The purpose of this trial is to evaluate the effects of combining task-oriented training with an electrical stimulation glove on hand function and dexterity in chronic stroke patients, compared to task-oriented training alone.

Study Design

This is a randomized controlled trial conducted at CMH Multan, Pakistan, over nine months. A total of 36 participants are enrolled, with 18 in each group. Patients are randomly assigned to either:

Intervention Group: Task-oriented training with an electrical stimulation glove.

Control Group: Task-oriented training only.

Eligibility Participants are men and women aged 40-60 years, at least six months after their first stroke, medically stable, and with adequate cognitive ability (Mini-Mental Scale score ≥24). Patients with recurrent stroke, seizures, pacemakers, or other neurological/orthopedic impairments are excluded.

Interventions

Task-Oriented Training (Control): Sessions include warm-up exercises, functional tasks such as pegboard placement, grasp-and-release of objects, writing or drawing, and simulated daily activities, followed by cool-down stretches.

Task-Oriented Training with Electrical Stimulation Glove (Intervention): Same activities as above, but performed while wearing the ESG. The glove delivers gentle electrical impulses to wrist and finger muscles during task performance, supporting active movement and sensory feedback.

Each session lasts approximately 60 minutes, including warm-up, 40 minutes of functional activities, and cool-down. The program runs three times per week for eight weeks.

Outcome Measures

Hand function and dexterity are evaluated before and after the intervention using standardized tools:

Wolf Functional Test (WFT): assesses the quality and speed of upper limb tasks.

Fugl-Meyer Assessment - Upper Extremity (FMA-U): evaluates motor recovery of the arm and hand.

Functional Dexterity Test (FDT): measures fine motor control and coordination.

Ethical Considerations Informed consent is obtained from all participants. Confidentiality and safety are maintained throughout the study. Participation is voluntary, and individuals may withdraw at any time without penalty.

ELIGIBILITY:
Inclusion Criteria:

* Patients after the six months of first stroke event (chronic stroke patient)
* Mini mental scale grade (24/above)
* Medically and neurologically stable condition
* No visual or auditory defects (Anderson & White, 2023)

Exclusion Criteria:

* Pre-existing arm impairment such as rheumatoid arthritis
* Cardiac pacemaker
* Patients with other neurological impairments
* Recurrent or progressive stroke
* Unconscious patients due to any other cause
* History of seizure within 2 years (Anderson & White, 2023)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Change in Upper Extremity Motor Function (Fugl-Meyer Assessment - Upper Extremity, FMA-U) | Baseline and 8 weeks post-intervention
  The Fugl-Meyer Assessment - Upper Extremity is a stroke-specific, performance-based scale that evaluates motor function, balance, sensation, and joint functioning. In this study, it is used to assess changes in upper limb motor recovery after intervention.

SECONDARY OUTCOMES:
Change in Functional Performance (Wolf Functional Test, WFT) | Baseline and 8 weeks post-intervention
  The Wolf Functional Test assesses upper extremity motor ability through timed and functional tasks such as lifting, reaching, and manipulating objects. It measures speed and quality of movement in stroke patients.
Change in Hand Dexterity (Functional Dexterity Test, FDT) | Baseline and 8 weeks post-intervention
  The Functional Dexterity Test evaluates fine motor control, coordination, and speed of finger movements required for daily activities. Lower scores reflect better dexterity.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackerley SJ, Byblow WD, Barber PA, MacDonald H, McIntyre-Robinson A, Stinear CM. Primed Physical Therapy Enhances Recovery of Upper Limb Function in Chronic Stroke Patients. Neurorehabil Neural Repair. 2016 May;30(4):339-48. doi: 10.1177/1545968315595285. Epub 2015 Jul 15. PMID 26180053
- [Background] Abo M, Kakuda W, Momosaki R, Harashima H, Kojima M, Watanabe S, Sato T, Yokoi A, Umemori T, Sasanuma J. Randomized, multicenter, comparative study of NEURO versus CIMT in poststroke patients with upper limb hemiparesis: the NEURO-VERIFY Study. Int J Stroke. 2014 Jul;9(5):607-12. doi: 10.1111/ijs.12100. Epub 2013 Sep 9. PMID 24015934